CLINICAL TRIAL: NCT05538494
Title: Short-term Effects on the Patellar Tendon After Low-load Blood-flow Restriction Training Versus High-load Conventional Training. Randomized Clinical Trial.
Brief Title: Effects on the Patellar Tendon After Low-load Blood Flow Restriction Training.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Alejandro Paricio Rufino, Physiotherapist, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TFMAON
Record Dates: First submitted 2022-08-26; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Patellar Tendinitis
Keywords: Patellar tendon; BFRT; vascular occlusion; Ultrasound; blood flow restriction training

STUDY DESIGN:
Intervention Model Description: The first group, which we will call the "BFR group", will be trained using low-load exercises with blood flow restriction. To the second group, which we will call "high load group", an exercise program with high loads will be applied.
Who Masked: Investigator
Masking Description: double blinding between investigator and study participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR group (Experimental): Training is applied to this group using low-load exercises with restriction of blood flow.
  Interventions: Other: BFR intervention
- High load group (Active Comparator): A program will be applied to this group of exercise with high loads as a method of treatment
  Interventions: Other: High load intervention

INTERVENTIONS:
Other: BFR intervention — Training is applied to this group using low-load exercises with restriction of blood flow. Based on the variables used by the major part of the protocols used in studies on the ERFS, the protocol that will be applied to this group will consist of the following parameters.
  * Training: 1 series of 30 repetitions followed by 3 series of 15 repetitions of squats
  * Rest between series: Duration of 45 seconds.
  * Workload: 30% of 1RM.
  * Cadence: 2 seconds for the concentric phase and 2 seconds for the eccentric phase (2:2).
  * Cuff pressure: The inflation pressure will be individualized for each individual.
  A pressure equivalent to 80% of the minimum pressure necessary for the total occlusion of the femoral artery.
  • Cuff placement: proximal quadriceps.
  Arms: BFR group
Other: High load intervention — A program will be applied to this group of exercise with high loads as a method of treatment in which the following will be applied parameters:
  * Training: 4 series of 12 repetitions of squats.
  * Rest between series: Duration 2 minutes.
  * Workload: 70% of 1RM.
  Arms: High load group

SUMMARY:
The main objective of this research project is to study the transient adaptations that occur in the tendon immediately after the object of training with low loads and blood flow restriction and to compare these adaptations with those derived from training with high loads, in order to thus helping to elucidate the complex existing framework regarding the effects of this training methodology on the tendon.

DETAILED DESCRIPTION:
Introduction: Nowadays, it is known that mechanical loading is essential to achieve tendon adaptations. So,if tendons are stimulated in the right way, positive changes will take part on the tendinous tissues increasing its capability to stand mechanical loading.In the last decade, low load blood flow restriction training has developed as an alternative methodto high load training, as some investigations have found a similar increase in force and hypertrophy between both training methods. Although, the evidence about tendon adaptations leading from low load blood flow restriction training is still very limited.Aim: The present study aims to study tendon temporary responses leading immediately after a low load blood flow restriction training and compare those adaptations with those leading from high load strength training.Design: A randomized case-control clinical trial will be conducted.Sample: The measurement of the sample size was done with theG*Power 3.1.5 program and was based on the time-by-group interaction of a mixed variance analysis (ANOVA). With two groups and three measurement moments. The final sample size was constituted by 84 subjectsMethods:The 84 participants will be randomly allocated in two groups: a) Low load blood flow restriction training (n=42); b) high load strength training (n=42). The low load blood flow restriction training group will perform a strength training with an intensity equivalent to 30% 1RM with an occlusion pressure of 80% on the total restriction pressure assessed individually, whilst the other group will train with a load equivalent of 80% 1RM. Patellar tendon characteristics will be studied as morphometry and densitometry parameters and microcirculation pre, post immediate intervention and 24 hourspost intervention.

ELIGIBILITY:
Inclusion Criteria:

* Physically active population (physical activity between 1 and 3 weekly sessions). With the final purpose to adjust the results to normality and refer to a general population.
* Subjects who have received the information sheet and have given their consent informed to participate in the study.

Exclusion Criteria:

* People who reproduce pain or symptomatology to the execution of the exercise of the treatment.
* People who have had symptoms in the last 2 months in the region below patellar
* Present musculoskeletal injuries or inability to perform the protocol experimental.
* Individuals with a training frequency equal to or greater than 5 sessions per week or that present a RM equal to or greater than 110kg. Since they do not fit a population and may affect the homogeneity of the sample.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-09-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate structural changes in the tendon through the use of ultrasound | Baseline
  Ultrasound will be used in order to collect the data of the images of each participants. Then, we will asses and compare possible changes in thickness, measured in cm, of each tendon before, after and 24 hour after the intervention.
To assest the echogenicity of each tendon by using software Fiji-Image J | Baseline
  A delimited area of 159x20 pixels inside the tendon structure will be selected. Then the program may classified all the pixels of each area on a gray scale of 255, resulting in an histogram of each tendon before, after and 24 hour after the intervention, measured in pixels in the gray scale.

OTHER OUTCOMES:
Evaluate the possible presence of micro vascularization of the patellar tendon through the visualization of the tendon structure with the doppler system of the ultrasound. | Baseline
  The Doppler mode of ultrasound will be used to observe and compare the presence of micro-vascularization inside the patellar tendon structure, before, immediately after and 24 hours after performing the intervention for each subject. The images where the doppler mode could detect some micro-vascularization may be assigned with ''Yes´´ and those which does not show any evidence of micro-vascularization ,may be assigned as ''no´´.

CONTACTS AND LOCATIONS:
Overall Officials: Néstro Ruíz Alberto, Physio, Principal Investigator — University of Alcala
Locations (1):
- University of Alcala, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] NEUBERGER A, PERRONE JC, SLACK HG. The relative metabolic inertia of tendon collagen in the rat. Biochem J. 1951 Jul;49(2):199-204. No abstract available. PMID 14858310
- [Background] Heinemeier KM, Kjaer M. In vivo investigation of tendon responses to mechanical loading. J Musculoskelet Neuronal Interact. 2011 Jun;11(2):115-23. PMID 21625048
- [Background] Onambele-Pearson GL, Pearson SJ. The magnitude and character of resistance-training-induced increase in tendon stiffness at old age is gender specific. Age (Dordr). 2012 Apr;34(2):427-38. doi: 10.1007/s11357-011-9248-y. Epub 2011 Apr 20. PMID 21505764
- [Background] Docking SI, Cook J. How do tendons adapt? Going beyond tissue responses to understand positive adaptation and pathology development: A narrative review. J Musculoskelet Neuronal Interact. 2019 Sep 1;19(3):300-310. PMID 31475937
- [Background] Magnusson SP, Narici MV, Maganaris CN, Kjaer M. Human tendon behaviour and adaptation, in vivo. J Physiol. 2008 Jan 1;586(1):71-81. doi: 10.1113/jphysiol.2007.139105. Epub 2007 Sep 13. PMID 17855761
- [Background] Kubo K, Ikebukuro T, Yaeshima K, Yata H, Tsunoda N, Kanehisa H. Effects of static and dynamic training on the stiffness and blood volume of tendon in vivo. J Appl Physiol (1985). 2009 Feb;106(2):412-7. doi: 10.1152/japplphysiol.91381.2008. Epub 2008 Dec 26. PMID 19112156
- [Background] Kubo K, Morimoto M, Komuro T, Yata H, Tsunoda N, Kanehisa H, Fukunaga T. Effects of plyometric and weight training on muscle-tendon complex and jump performance. Med Sci Sports Exerc. 2007 Oct;39(10):1801-10. doi: 10.1249/mss.0b013e31813e630a. PMID 17909408
- [Background] Grigg NL, Wearing SC, Smeathers JE. Eccentric calf muscle exercise produces a greater acute reduction in Achilles tendon thickness than concentric exercise. Br J Sports Med. 2009 Apr;43(4):280-3. doi: 10.1136/bjsm.2008.053165. Epub 2008 Nov 19. PMID 19019906
- [Background] Iwanuma S, Akagi R, Kurihara T, Ikegawa S, Kanehisa H, Fukunaga T, Kawakami Y. Longitudinal and transverse deformation of human Achilles tendon induced by isometric plantar flexion at different intensities. J Appl Physiol (1985). 2011 Jun;110(6):1615-21. doi: 10.1152/japplphysiol.00776.2010. Epub 2011 Mar 17. PMID 21415176
- [Background] Cook JL, Purdam CR. Is tendon pathology a continuum? A pathology model to explain the clinical presentation of load-induced tendinopathy. Br J Sports Med. 2009 Jun;43(6):409-16. doi: 10.1136/bjsm.2008.051193. Epub 2008 Sep 23. PMID 18812414
- [Background] Syha R, Springer F, Grozinger G, Wurslin C, Ipach I, Ketelsen D, Schabel C, Gebhard H, Hein T, Martirosian P, Schick F, Claussen CD, Grosse U. Short-term exercise-induced changes in hydration state of healthy Achilles tendons can be visualized by effects of off-resonant radiofrequency saturation in a three-dimensional ultrashort echo time MRI sequence applied at 3 Tesla. J Magn Reson Imaging. 2014 Dec;40(6):1400-7. doi: 10.1002/jmri.24488. Epub 2013 Nov 8. PMID 24214925
- [Background] Scott BR, Loenneke JP, Slattery KM, Dascombe BJ. Exercise with blood flow restriction: an updated evidence-based approach for enhanced muscular development. Sports Med. 2015 Mar;45(3):313-25. doi: 10.1007/s40279-014-0288-1. PMID 25430600
- [Background] Chulvi-Medrano I, Picon-Martinez M, Cortell-Tormo JM, Tortosa-Martinez J, Alonso-Aubin DA, Alakhdar Y. Different Time Course of Recovery in Achilles Tendon Thickness After Low-Load Resistance Training With and Without Blood Flow Restriction. J Sport Rehabil. 2020 Jul 27;30(2):300-305. doi: 10.1123/jsr.2019-0403. PMID 32717720
- [Background] Hullfish TJ, Baxter JR. A Reliable Method for Quantification of Tendon Structure Using B-Mode Ultrasound. J Ultrasound Med. 2018 Oct;37(10):2419-2424. doi: 10.1002/jum.14592. Epub 2018 Mar 25. PMID 29574900
- [Background] Cook JL, Khan KM, Harcourt PR, Kiss ZS, Fehrmann MW, Griffiths L, Wark JD. Patellar tendon ultrasonography in asymptomatic active athletes reveals hypoechoic regions: a study of 320 tendons. Victorian Institute of Sport Tendon Study Group. Clin J Sport Med. 1998 Apr;8(2):73-7. doi: 10.1097/00042752-199804000-00001. PMID 9641432
- [Background] Rios-Diaz J, de Groot Ferrando A, Martinez-Paya JJ, del Bano Aledo ME. [Reliability and reproducibility of a morpho-textural image analysis method over a patellar ligament ultrasonography]. Reumatol Clin. 2010 Nov-Dec;6(6):278-84. doi: 10.1016/j.reuma.2010.01.008. Epub 2010 May 13. Spanish. PMID 21794733
- [Background] Hansen P, Bojsen-Moller J, Aagaard P, Kjaer M, Magnusson SP. Mechanical properties of the human patellar tendon, in vivo. Clin Biomech (Bristol). 2006 Jan;21(1):54-8. doi: 10.1016/j.clinbiomech.2005.07.008. Epub 2005 Sep 23. PMID 16183183
- [Background] Martínez Payá JJ, Ríos Díaz J, Baño Aledo, María Elena del. El análisis textural mediante las matrices de co-ocurrencia (GLCM) sobre la imagen ecográfica del tendón rotuliano es de utilidad para la detección de cambios histológicos tras un entrenamiento con plataforma de vibración. Cultura, ciencia y deporte 2009;4(11):91-102.
- [Background] Cobos-Carbo A, Augustovski F. [CONSORT 2010 Declaration: updated guideline for reporting parallel group randomised trials]. Med Clin (Barc). 2011 Jul 23;137(5):213-5. doi: 10.1016/j.medcli.2010.09.034. Epub 2011 Jan 15. No abstract available. Spanish. PMID 21239025
- [Background] Abe T, Yasuda T, Midorikawa T, Sato Y, CF K, Inoue K, et al. Skeletal muscle size and circulating IGF-1 are increased after two weeks of twice daily "KAATSU" resistance training. International Journal of KAATSU Training Research 2005;1(1):6-12.
- [Background] Risch L, Mayer F, Cassel M. Doppler Flow Response Following Running Exercise Differs Between Healthy and Tendinopathic Achilles Tendons. Front Physiol. 2021 Mar 23;12:650507. doi: 10.3389/fphys.2021.650507. eCollection 2021. PMID 33833692
- [Background] Balsalobre-Fernandez C, Marchante D, Munoz-Lopez M, Jimenez SL. Validity and reliability of a novel iPhone app for the measurement of barbell velocity and 1RM on the bench-press exercise. J Sports Sci. 2018 Jan;36(1):64-70. doi: 10.1080/02640414.2017.1280610. Epub 2017 Jan 18. PMID 28097928
- [Background] Giles L, Webster KE, McClelland J, Cook JL. Quadriceps strengthening with and without blood flow restriction in the treatment of patellofemoral pain: a double-blind randomised trial. Br J Sports Med. 2017 Dec;51(23):1688-1694. doi: 10.1136/bjsports-2016-096329. Epub 2017 May 12. PMID 28500081
- [Background] Moisés Picón Martínez. Efectos agudos del entrenamiento con restricción del flujo sanguíneo sobre el tendón, la respuesta cardiovascular y la respuesta muscular Universitat d'Alacant - Universidad de Alicante; 2018.
- [Background] Ladlow P, Coppack RJ, Dharm-Datta S, Conway D, Sellon E, Patterson SD, Bennett AN. Low-Load Resistance Training With Blood Flow Restriction Improves Clinical Outcomes in Musculoskeletal Rehabilitation: A Single-Blind Randomized Controlled Trial. Front Physiol. 2018 Sep 10;9:1269. doi: 10.3389/fphys.2018.01269. eCollection 2018. PMID 30246795